CLINICAL TRIAL: NCT04479150
Title: Postoperative Complications and Mortality of Patients Submited to Emergency Digestive Surgery During the COVID-19 Pandemic (COVIDCIR Study): a Multicenter Cohorts' Study Protocol
Brief Title: Complications and Mortality Following Emergency Digestive Surgery During the COVID-19 Pandemic
Acronym: COVIDCIR
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Javier Osorio, Javier Osorio, Hospital Universitari de Bellvitge
Other Study IDs: COVIDCIR
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Surgery--Complications
Keywords: Covid19; Emergency surgery; Postoperative complications; Postoperative mortality
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pandemic Covid-positive cohort: All Covid-positive patients operated on for emergency digestive pathology from March, 1st 2020 to June, 30th 2020
- Pandemic Covid-negative cohort: All Covid-negative patients operated on for emergency digestive pathology from March, 1st 2020 to June, 30th 2020
- Control cohort: Pre-pandemic cohort: all patients operated on for emergency digestive pathology from March, 1st 2020 to June, 30th 2019.

SUMMARY:
A multi-centre, observational cohort study will be carried out in consecutive patients operated on for urgent digestive pathology. Two cohorts will be defined: the 'pandemic' cohort, which will include all patients [COVID-19-positive or negative] operated on for emergency digestive pathology during the months of March to June 2020; and the control cohort, which will include all patients operated on for emergency digestive pathology during the months of March to June 2019.

Information will be gathered on demographic characteristics, clinical and analytical parameters, scores on the usual risk scales for quality management in a General Surgery service (POSSUM, P-POSSUM and LUCENTUM scores), prognostic factors applicable to all patients, specific factors for patients infected with SARS-CoV-2, complications and postoperative mortality (at 30 and 90 postoperative days). In the pandemic cohort it will be detailed whether or not the patient was infected with SARS-CoV-2.

The main objective will be to determine the incidence of postoperative complications and mortality. This variable will be analysed in the "full analysis set" population. Secondary objective will be to develop a specific postoperative risk propensity model for SARS-CoV-2 infected patients.

DETAILED DESCRIPTION:
COVIDCIR is an observational, multicenter, cohorts' study of patients undergoing emergency/urgent gastrointestinal surgery during the period of maximum impact of the COVID-19 pandemic in Spain (from March 1st to June 30th, 2020).

The study conforms to the stipulations of the Declaration of Helsinki. The protocol was approved by the local Institutional Review Board (Ethics and Clinical Investigation Committee) and a waiver for written informed consent was given. The level of protection of confidentiality, in terms of protection of personal data as required by Spanish Law (LOPD 3/2018), was also ensured.

A total of 30 surgical teams from different Spanish hospitals have been proposed as participants in this study, which has been coordinated by the Department of General and Digestive Surgery of Bellvitge University Hospital (L'Hospitalet del Llobregat, Barcelona, Spain). All hospitals participating are from Spain, with different surgical capabilities.

Patients operated on for emergency/urgent gastrointestinal surgery constitute the target population.

Inclusion criteria: ≥18 years, both genders, and operated on for urgent/emergency gastrointestinal pathology.

Exclusion criteria: patients who have undergone a scheduled surgical intervention or patients operated on by a service other than General and Digestive Surgery.

Three cohorts will be defined:

Cohort 1: Covid-19-positive (infected by SARS-CoV-2) patients who required emergency/urgent gastrointestinal surgery from March 1st to June 30th, 2020 Cohort 2: Covid-19-negative (not infected by SARS-CoV-2)patients who required emergency/urgent gastrointestinal surgery from March 1st to June 30th, 2020.

Cohort 3: Consecutive patients who required emergency/urgent gastrointestinal surgery from March 1st to June 30th, 2019 (control cohort of a "pre-pandemic" period, all patients Covid-19-negative).

Primary outcome is 30-day postoperative mortality. Secondary variables are 90-day mortality, postoperative complications, severa complications (graded as Clavien-Dindo score >= IIIA), and length of stay.

Main variables related to postoperative mortality and complications will be: Age, comorbidities, ASA score, type of surgical pathology, type of performed surgery, POSSUM score, P-POSSUM score, LUCENTUM score and specific analitic parameters for Covid-19 patients.

Baseline characteristics will be summarized using standard descriptive statistics, and a descriptive and exploratory comparative analysis between cohorts will be carried out.

The cumulative incidence of mortality (and its 95% confident interval) and the incidence of morbidity (and its 95% confident interval) at 30 and 90 days will be estimated by SARS-CoV-2 infection status (cohort 1) and in the control groups (cohorts 2 and 3).

To minimize the selection bias effect of potential confounders, propensity scores will be estimated using a multinomial model to estimate the probability that subjects were SARS-CoV-2-positive, SARS-CoV-2-negative. Then, subjects will be matched using the propensity score. After matching, to identify imbalance between groups, the standardized mean difference will be estimated and plotted. In the matched sample, the cumulative incidence of mortality (and its 95% confidence interval) and the incidence of morbidity (and its 95% confidence interval) at 30 and 90 days will be compared using a generalized linear model with a binomial distribution and a logarithm link function. Those variables that remain imbalance between groups after matching would be added to the model with an adjusting purpose.

A generalized linear model with a binomial distribution and a logarithm link function will be used to estimate relative risk as a measure to indentify prognostic factors associated with 30 and 90 days mortality and morbidity incidences. Five predictive scores of postoperative complications and/or mortality will be calculated: POSSUM-mortality, POSSUM-complications, P-POSSUM, LUCENTUM-logistic regression and LUCENTUM-CHAID. Their applicability on the complications and/or mortality prediction in COVID-19 pandemic will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥18 years, both genders, and operated on for urgent/emergency gastrointestinal pathology.

Exclusion Criteria:

* Patients who have undergone a scheduled surgical intervention or patients operated on by a service other than General and Digestive Surgery.
* Patients < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for emergency/urgent gastrointestinal surgery constitute the target population.
Sampling Method: Non-Probability Sample
Enrollment: 5307 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days post-surgery
  Mortality for any cause at 30 days after urgent gastrointestinal surgery.

SECONDARY OUTCOMES:
90-day mortality | 90 days post-surgery
  Mortality for any cause within 90 days of surgery
Postoperative complications | 30 days post-surgery
  Postoperative complications within 30 days of surgery: classic postoperative complications, typical complications after digestive surgery and/or complications specifically associated with the evolution of COVID-19
Severe complications | 30 days post-surgery
  Postoperative complications within 30 days of surgery graded as equal or superior to IIIA grade according to the Clavien-Dindo classification
Lenght of stay | 90 days post-surgery
  Number of days of hospital stay from the day of admission to the date of hospital discharge or death

CONTACTS AND LOCATIONS:
Overall Officials: Javier Osorio, MD, PhD, Principal Investigator — Hospital Universitary de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Osorio J, Madrazo Z, Videla S, Sainz B, Rodriguez-Gonzalez A, Campos A, Santamaria M, Pelegrina A, Gonzalez-Serrano C, Aldeano A, Sarriugarte A, Gomez-Diaz CJ, Ruiz-Luna D, Garcia-Ruiz-de-Gordejuela A, Gomez-Gavara C, Gil-Barrionuevo M, Vila M, Clavell A, Campillo B, Millan L, Olona C, Sanchez-Cordero S, Medrano R, Lopez-Arevalo CA, Perez-Romero N, Artigau E, Calle M, Echenagusia V, Otero A, Tebe C, Pallares N, Biondo S; COVID-CIR Collaborative Group Members of the COVID-CIR Collaborative Group. Analysis of outcomes of emergency general and gastrointestinal surgery during the COVID-19 pandemic. Br J Surg. 2021 Dec 1;108(12):1438-1447. doi: 10.1093/bjs/znab299. PMID 34535796
- [Derived] Madrazo Z, Osorio J, Otero A, Biondo S, Videla S; on behalf of The COVID-CIR Collaborative Group. Postoperative complications and mortality following emergency digestive surgery during the COVID-19 pandemic: A multicenter collaborative retrospective cohort study protocol (COVID-CIR). Medicine (Baltimore). 2021 Feb 5;100(5):e24409. doi: 10.1097/MD.0000000000024409. PMID 33592888